CLINICAL TRIAL: NCT05506813
Title: Comparative Effects of Cognitive and Motor Dual Task Training on Balance and Quality Of Life in Parkinson's Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: REC/RCR & AHS/21/0256
Record Dates: First submitted 2022-08-17; First posted 2022-08-18 (Actual); Last update posted 2022-11-09 (Actual); Status verified 2022-11

CONDITIONS: Parkinson Disease; Balance; Distorted; Postural; Defect
Keywords: Parkinson Disease; Balance; Distorted; Postural; Defect
MeSH Terms: conditions — Parkinson Disease | interventions — Cognitive Training

STUDY DESIGN:
Intervention Model Description: total 20 Participants will be divided in two groups. In group A patients will receive cognitive training along with conventional therapy. while in Group B Participants will receive motor dual task training along with conventional therapy.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- experimental group (Experimental): cognitive training and conventional training
  Interventions: Other: cognitive training and conventional training
- control group (Active Comparator): motor dual task training and conventional training
  Interventions: Other: motor dual task training along with conventional therapy

INTERVENTIONS:
Other: cognitive training and conventional training — cognitive training along with conventional therapy
  Arms: experimental group
Other: motor dual task training along with conventional therapy — motor dual task training along with conventional therapy
  Arms: control group

SUMMARY:
To Compare Effects of Cognitive and Motor Dual Task Training on Balance and Quality Of Life in Parkinson's Patients

DETAILED DESCRIPTION:
This study will be conducted to compare the Comparative Effect of Cognitive and Motor Dual Task Training on Balance and Quality Of Life in Parkinson's Patients. total 20 Patients will be recruited according to the inclusion criteria and data will be collected from the Riphah Rehabilitation center Lahore, Muhammadi Medical trust hospital Lahore. Time Up and Go test (TUG) Parkinsons disease Questionnaire 39 (PDQ-39) will be used as data collection tool. To assess the balance and quality of life in parkinson's patients. Patients will be allocated to intervention group by randomization. After approval from ethical committee, data collection will be started and informed consent will be taken from all patients

ELIGIBILITY:
Inclusion Criteria:

* A stage I-II-III Hoehn and Yahr scale consultant neurologist's diagnosis of Parkinson's disease
* A stable medication schedule both before and during the trial period
* can walk without assistive aid

Exclusion Criteria:

* Other neurological conditions in additions to Parkinson's disease such as CVA, Head injuries, Trauma
* Any Musculoskeletal condition e.g., total knee replacement surgery and rheumatoid arthritis
* Sensory impairments (vestibular dysfunctions)

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2022-08-20 (Actual); Study Completion 2022-08-20 (Actual)

PRIMARY OUTCOMES:
time up and go test | 9 months
  In time up and go test instruct patient stand up and then walking 3 meters far then rotate and come back. Therapist noted the whole procedure time
Parkinson Disease Questionnaire-39 (PDQ-39). | 9 months
  Parkinson Disease Questionnaire-39 (PDQ-39).The tool carried out 39 items. The tool carried out 39 items. For each domain, five answer shows that every part score is 0 (good) to 100 (critical). Decreased scores showed better quality of life

CONTACTS AND LOCATIONS:
Overall Officials: Zeest Hashmi, MSNMPT, Principal Investigator — Riphah International University
Locations (1):
- Riphah International University, Islamabad, Fedral, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bordignon A, Devita M, Sergi G, Coin A. "Cerebellar cognitive reserve": a possible further area of investigation. Aging Clin Exp Res. 2021 Oct;33(10):2883-2886. doi: 10.1007/s40520-021-01795-1. Epub 2021 Feb 17. No abstract available. PMID 33595777
- [Background] Onder H, Ozyurek O. The impact of distinct cognitive dual-tasks on gait in Parkinson's disease and the associations with the clinical features of Parkinson's disease. Neurol Sci. 2021 Jul;42(7):2775-2783. doi: 10.1007/s10072-020-04874-9. Epub 2020 Nov 4. PMID 33150515
- [Background] Bouscary A, Quessada C, Rene F, Spedding M, Turner BJ, Henriques A, Ngo ST, Loeffler JP. Sphingolipids metabolism alteration in the central nervous system: Amyotrophic lateral sclerosis (ALS) and other neurodegenerative diseases. Semin Cell Dev Biol. 2021 Apr;112:82-91. doi: 10.1016/j.semcdb.2020.10.008. Epub 2020 Nov 5. PMID 33160824